CLINICAL TRIAL: NCT01636128
Title: A Phase 2 Urinary Biomarker Study of Polyamine Inhibition With Sulindac and Difluoromethylornithine (DFMO)
Brief Title: Urinary Biomarker Study With Sulindac and Difluoromethylornithine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding and staffing
Sponsor: Cancer Prevention Pharmaceuticals, Inc. (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Patricia Thompson-Carino, Associate Professor, Cellular and Molecular Medicine, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UA-UB-101
Record Dates: First submitted 2012-07-02; First posted 2012-07-10 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Focus of Study: Drug Response Biomarkers, Chemoprevention, Neoplasms
Keywords: Urinary; biomarkers; DFMO; sulindac
MeSH Terms: conditions — Neoplasms | interventions — Eflornithine; Sulindac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulindac first (Treatment Sequence B) (Experimental): Sulindac alone, washout, DFMO alone, then combination of sulindac and DFMO
  Interventions: Drug: difluoromethylornithine; Drug: Sulindac
- DFMO first (Treatment Sequence A) (Experimental): DFMO alone, followed by washout, sulindac alone, then combination of DFMO and sulindac
  Interventions: Drug: difluoromethylornithine; Drug: Sulindac

INTERVENTIONS:
Drug: difluoromethylornithine — 500 mg oral for 14 days, combined with sulindac for 15 days
  Other Names: DFMO, eflornithine
Drug: Sulindac — 150 mg oral for 15 days, combined with DFMO for 14 days

SUMMARY:
The purpose of this study is to determine the effects of 2 drugs (sulindac and Difluoromethylornithine (DFMO)) either alone or in combination on biomarkers found in urine.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years
* Fluent in English
* PS 0 ECOG
* Must be able to discontinue the use of aspirin, aspirin containing products, and other non-steroidal anti-inflammatory agents for the duration of the study agent administration period
* Negative fecal occult blood test
* Hemoglobin > 10g/dl, WBC must be >4,000 mm3, platelets must be > 100,000/mm3
* Serum creatinine must be < 1.5 m/dl
* Serum bilirubin must be < 2.0 mg/dl, AST and ALT must be < 1.5x upper limit of normal range
* Female participants must be postmenopausal (at least 1 year since the last menstrual period), surgically sterilized, or willing to use an effective birth control method (e.g., hormonal contraceptive, oral contraceptives, intrauterine device, diaphragm with spermicide, or abstinence) for the duration of the study. Male subjects must use an effective method of birth control throughout the duration of the study and should not impregnate a female.
* Females of childbearing potential must have a negative serum pregnancy test prior to the start of study medication.
* Able to give signed, written informed consent

Exclusion Criteria:

* Requires corticosteroids or nonsteroidal anti-inflammatory agents
* Individuals who are immunosuppressed by virtue of medication or disease. This includes participants known to have AIDS, subjects taking oral steroids, and subjects on immunosuppressants/immunomodulators (cyclosporine, chemotherapeutic agents, or biologic therapy)
* Current use of phenytoin or sulfonamides
* Current or recent (within 3 months) use of coumadin or other systemic anticoagulants.
* Frequently, chronic or moderate/severe gastric complaints. Upper gastrointestinal problems requiring prescription or nonprescription medical remedies for symptoms of heartburn, dyspepsia, nausea, or abdominal pain > once per week on average
* History of peptic ulcer, occult or gross intestinal bleeding
* Known intercurrent illness, including but no limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, renal disease, liver disease, ongoing or active infection, psychiatric illness, or other situations that would limit compliance or interfere with the ability to comply with the study regimen.
* History of bleeding or clotting disorders
* Individuals with seizures or history of seizures
* History of abnormal wound healing or repair, or conditions that predisposes to the same including diabetes
* Unwilling or unable to limit alcohol consumption to 2-3 servings per week during the study period (12oz beer, 1 oz per alcoholic beverage, 6 oz per wine)
* Individuals enrolled in or who plan to enroll in a clinical intervention trial. There must be a 30 day period between completing a previous study and enrolling in this study.
* Pregnant or lactating women
* Prior DFMO exposure
* History of allergic reaction (e.g., urticaria, asthma, rhinitis) or gastric intolerance attributed to NSAIDs

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Measure intra-subject urine N1-monoacetylspermidine and dcSAM variability during the pre-drug phase | Week 1-Week 2
  Measure initial variability in levels of urinary biomarkers prior to initiation of drug treatment. Three blood draws over the first 14 days will be used to assess baseline variability.
Determine dcSAM content of urine after 14 days of 500mg DFMO daily alone | Week 4
  Measure urinary biomarker dcSAM after 14 days of single agent DFMO. Measure urinary biomarker dcSAM after 14 days of single agent DFMO for treatment arm where DFMO alone is started week 2 (Treatment sequence A).
Determine N1-monoacetylspermidine content of urine after 14 days plus 1 day of 150 mg sulindac alone | Week 4
  Measure urinary biomarker dcSAM after 14 days of single agent sulindac. Measure urinary biomarker dcSAM after 14 days of single agent sulindac for treatment arm where sulindac alone is started week 2 (Treatment sequence B).
Determine dcSAM and N1-monoacetylspermidine content of urine after 14 days of 150 mg sulindac daily combined with DFMO at 500 mg/day | Week 20
Determine dcSAM content of urine after 14 days of 500mg DFMO daily alone | Week 12
  Measure urinary biomarker dcSAM after 14 days of single agent DFMO for treatment arm where DFMO alone is started week 10 (Treatment sequence B)
Determine N1-monoacetylspermidine content of urine after 14 days plus 1 day of 150 mg sulindac alone | Week 12
  Measure urinary biomarker dcSAM after 14 days of single agent sulindac. Measure urinary biomarker dcSAM after 14 days of single agent sulindac for treatment arm where sulindac alone is stated week 10 (Treatment sequence A).

SECONDARY OUTCOMES:
Determine if 2 weeks is sufficient time for dcSAM levels and N1-monoacetylspermidine content of urine to recover after stopping DFMO and sulindac | Week 22
Determine the length of time it takes for sulindac or DFMO to induce measurable changes in biomarker content of urine | Week 3-Week 25
Explore the effect of dietary intake of polyamine measured using the Arizona Food Frequency Questionnaire | Week 1-25
  Quantitate dietary polyamine levels over the course of the study and evaluate the effects on biomarkers evaluated in the primary outcome measures.